CLINICAL TRIAL: NCT07015424
Title: Prospective, Randomized Clinical Study Evaluating Transoral Outlet Reduction (TORe) and Lifestyle Modification for Patients With Weight Regain Following Roux-en-Y Gastric Bypass
Brief Title: Randomized Study on Transoral Outlet Reduction and Lifestyle Changes for Weight Regain After Gastric Bypass
Acronym: REIGNITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7220
Record Dates: First submitted 2025-05-21; First posted 2025-06-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Weight Regain; Weight Loss
Keywords: TORe; OverStitch
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TORe and Lifestyle Modification Arm (Active Comparator): Subjects will receive a TORe procedure and intensive lifestyle modification throughout the study
  Interventions: Device: TORe with OverStitch; Behavioral: Intensive lifestyle modification
- Lifestyle Modification Arm (Active Comparator): Subjects will receive intensive lifestyle modification throughout the study. At 6 months post enrollment, subjects will be eligible to receive a TORe procedure.
  Interventions: Behavioral: Intensive lifestyle modification

INTERVENTIONS:
Device: TORe with OverStitch — Transoral Outlet Reduction with OverStitch Endoscopic Suturing System
  Arms: TORe and Lifestyle Modification Arm
Behavioral: Intensive lifestyle modification — Intensive lifestyle modification program consists of the following: well-balanced calorie-restrictive diet, incorporation of exercise and coaching on lifestyle changes. The program should include personal discussions and goals designed and overseen by the treating physician, obesity management professional or dietician.

SUMMARY:
The goal of this clinical trial is to evaluate weight loss with TORe and intensive lifestyle modification versus intensive lifestyle modification alone in subjects who have regained weight following a Roux-en-Y gastric bypass.

Participants will randomized 2:1. Those randomized to the TORe arm will receive a TORe procedure and intensive lifestyle modification which consists of a well-balanced calorie restrictive diet, incorporation of exercise and coaching on lifestyle discussion. Participants randomized the lifestyle modification alone arm will be eligible to receive a TORe procedure at 6 months post enrollment. Total follow up will be 24 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Experiencing weight regain (≥ 20% weight from nadir) after achieving clinically successful weight loss.
* Willing to have a TORe procedure for the treatment of weight regain.
* BMI between 30 and 50 kg/m2, inclusive.
* GJA diameter ≥ 20 mm, confirmed either during a
* Screening EGD completed ≤ 60 days from study procedure or
* EGD performed immediately prior to the TORe procedure.
* Anatomically accepting of the procedure, including a pouch size that will not require reduction at the time of treatment (pouch that is shorter than 6 cm in length).
* Agrees not to take additional over the counter or prescribed weight loss supplements / medications (including incretins) during the first 6 months of the study.
* Is on a stable dose of anti-diabetic medication for three months with no anticipated changes during the first 6 months of the study.
* Agrees to the follow-up requirements of the study and is able to read, understand, and sign a written Informed Consent Form to participate in the study.
* Meets the indications for TORe procedure with OverStitch™ Endoscopic Suturing System.

Exclusion Criteria:

* Current use or use within the three months prior to the baseline visit of over the counter or prescribed weight loss supplements / medications (including incretins).
* Current or planned management of Type 2 Diabetes with incretin medications.
* Inability or unwillingness to comply with assigned treatment or protocol requirements related to visits.
* Investigator's medical judgement that the subject is not a candidate for the TORe procedure.
* Current pregnancy confirmed by site standard of care or planned pregnancy or breastfeeding in the next two years.
* Vulnerable subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Total Body Weight Loss | 6 Months post enrollment
  The percent TBWL that subjects achieve at 6 months post-randomization

SECONDARY OUTCOMES:
Clinically significant weight loss | 6, 12 and 24 months post enrollment
  The rate of subjects that achieve clinically significant weight loss (i.e. responders) at 6 months. Clinically significant weight loss is defined as ≥ 10% TBWL.
Percent TBWL at each visit | 6 months post enrollment and through end of study
  Percent TBWL at each visit
Change in A1C | 6, 12, 18, and 24 months post enrollment
  Change in Hemoglobin A1C from baseline
Change in Insulin | 6, 12, 18, and 24 months post enrollment
  Change in Insulin from baseline
Change in Fasting Glucose | 6, 12, 18, and 24 months post enrollment
  Change in Fasting Glucose from baseline
Change in Cholesterol | 6, 12, 18, and 24 months post enrollment
  Change in Total Cholesterol from baseline
Change in LDL | 6, 12, 18, and 24 months post enrollment
  Change in LDL from baseline
Change in HDL | 6, 12, 18, and 24 months post enrollment
  Change in HDL from baseline
Change in Triglycerides | 6, 12, 18, and 24 months post enrollment
  Change in Triglycerides from baseline
Change in Alanine transaminase (ALT) | 6, 12, 18, and 24 months post enrollment
  Change in ALT from baseline
Change in Alkaline phosphatase (ALP) | 6, 12, 18, and 24 months post enrollment
  Change in ALP from baseline
Change in Aspartate aminotransferase (AST) | 6, 12, 18, and 24 months post enrollment
  Change in AST from baseline
Reduction in Medications for Type 2 diabetes | 6, 12, 18 and 24 months post enrollment
  Reduction in Type 2 diabetes medication dose and frequency from Baseline
Reduction in Hypertension Medication | 6, 12, 18 and 24 months post enrollment
  Reduction in hypertension medication dose and frequency from Baseline
Reduction in cholesterol medication | 6, 12, 18 and 24 months post enrollment
  Reduction in cholesterol medication dose and frequency from Baseline
Reduction in medications for dumping syndrome | 6, 12, 18 and 24 months post enrollment
  Reduction in dumping syndrome medication dose and frequency from Baseline
Number of device and procedure-related Adverse Events (AEs) and Serious Adverse Events (SAEs) | From enrollment through 24 months (study completion)
  Continuous assessment of safety of TORe by summarizing the occurrence of device and procedure-related Adverse Events (AEs) and Serious Adverse Events (SAEs) at all visits and overall.
Change in Impact of Weight on Quality of Life (IWQOL LITE-CT) Quality of Life Questionnaire | 6, 12, 18, and 24 months post enrollment
  Change in IWQOL LITE-CT scores from baseline
Change in 36-Item Short Form Survey (SF-36) Quality of Life Questionnaire | 6, 12, 18, and 24 months post enrollment
  Change in SF-36 Questionnaire scores from baseline
Change in Sigstad Score | 6, 12, 18, and 24 months post enrollment
  Change in Sigstad score from baseline

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Hoag Memorial Hospital, Irvine, California
  - Stanford University Medical Center, Stanford, California
  - Mayo Clinic, Jacksonville, Florida
  - Orlando Health Inc, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic Foundation, Rochester, Minnesota
  - NYU Grossman School of Medicine, New York, New York
  - University of Texas Houston Health Science Center, Houston, Texas